CLINICAL TRIAL: NCT06816693
Title: Feasibility Study of a Mobile Application (App)-Based Tele-cardiac Rehabilitation (Tele-CR) Program for Patients With Coronary Heart Disease (CHD): Mixed Methods
Brief Title: Exploratory Study of the Usability, Feasibility, and Perception for Tele-cardiac Rehabilitation (Tele-CR) Program
Acronym: Tele-CR
Status: Enrolling by invitation | Type: Observational
Sponsor: Chang Gung University of Science and Technology (Other)
Collaborators: Chang Gung University (Other); Chang Gung Memorial Hospital (Other); National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 202301928B0
Record Dates: First submitted 2025-01-22; First posted 2025-02-10 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-02

CONDITIONS: Coronary Heart Disease; Coronary Arterial Disease (CAD)
Keywords: coronary heart disease; cardiac rehabilitation; telemedicine; mobile health
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- A tele-CR program was implemented for all participants: A 12 weeks tele-CR program was implemented for all participants.
  Interventions: Behavioral: tele-CR program

INTERVENTIONS:
Behavioral: tele-CR program — Following the completion of basic characteristics assessment prior to discharge, a 12 weeks tele-CR program was implemented for all participants. The tele-CR program is divided into three parts: motivational interview, App delivery, and self-management and tracking. The motivational interviewing during hospitalization, which involved evaluating individual risk factors, setting behavioral goals, and providing training on the installation and operation of the tele-CR App (approximately 30-60 minutes per session). After discharge, the researchers monitored App usage and conducted four follow-up sessions via LINE or telephone at 1, 4, 8, and 12 weeks post-discharge. These follow-ups, lasting approximately 5-15 minutes each, aimed to assess patients' living conditions, resolve any issues promptly, and provide encouragement or praise based on their engagement with the App.

SUMMARY:
The goal of this mixed prospective observational and qualitative studies is to evaluate the usability of a newly developed application (App) and the feasibility and perception of a 12 weeks tele-cardiac rehabilitation (tele-CR) program. The main question it aims to answer is: Does tele-CR program intervention a acceptance feasibility in coronary heart disease patients? The findings will guide subsequent intervention design studies.

DETAILED DESCRIPTION:
CHD is one of the leading causes of death in worldwide and Taiwan. While tele-CR holds the potential to reduce the readmission and improve the quality of life of patients with CHD, there is currently a paucity of research on this technology in Taiwan. Currently, traditional cardiac rehabilitation is the main method in Taiwan. However, the problem of under-usage in traditional cardiac rehabilitation after discharge persists. Literature shows that tele-CR may be a safe and effective supplement or alternative strategy. Therefore, we plan to develop a feasible tele-CR Program to optimize the quality of continuing care for CHD patients. The purpose of this study includes: 1. Develop App and management platform. 2. Understand the usability of the App in the 4th and 12th weeks. 3. Understand tele-CR program recruitment rates. 4. To understand the engagement rate of tele-CR program in the 1st, 4th, 8th and 12th weeks. 5. To understand the retention rate of tele-CR program at 1, 4, 8 and 12 weeks. 6. Understand the experience of receiving tele-CR program (qualitative).

A mixed methods approach will be used, including prospective observational and qualitative research designs. The study will be conducted in the cardiology ward of a medical center in the Northern District. A purposive sampling of patients admitted to the hospital with a primary diagnosis of CHD will be conducted. We estimate that we will recruit 45 cases (quantitative).

This study was reviewed and approved by the Institutional Review Board (IRB) of the study hospital. Research assistants provided detailed explanations of the study's purpose and procedures to potential participants who met the inclusion criteria. Any questions or concerns raised by the participants were addressed before obtaining written informed consent. Data collection was conducted only after consent was secured. Questionnaire data were obtained either through self-administration or via research assistants, who posed the questions individually based on the participants' needs. All data collection took place in a quiet and undisturbed environment to ensure accuracy and comfort.

All participants will undergo tele-CR for 12 weeks after completing the basic characteristics assessment. After discharge, the researchers monitored App usage and conducted four follow-up sessions via LINE or telephone at 1, 4, 8, and 12 weeks post-discharge. These follow-ups, lasting approximately 5-15 minutes each, aimed to assess patients' living conditions, resolve any issues promptly, and provide encouragement or praise based on their engagement with the App.

To evaluate the App's acceptance and usability, the Technology Acceptance Model Scale (TAMS) and System Usability Scale (SUS) were administered during the 4th and 12th weeks. Data collection methods included telephone or in-person sessions, allowing participants to complete the questionnaires either independently or through a question-and-answer format according to their preference. At the 8th-week telephone follow-up, participants were invited to engage in one-on-one semi-structured in-depth interviews. These interviews were scheduled at the participants' convenience and conducted in a quiet, private setting. With participants' consent, the interviews were audio-recorded, and researchers documented non-verbal behaviors for additional insights. If participants could not be reached via telephone, follow-up appointments were coordinated during outpatient visits to ensure data integrity and minimize participant attrition or data discrepancies. This approach was designed to enhance the reliability of the study findings. The recruitment, engagement, and retention rates will also be calculated. Data analysis will be performed using SPSS 26.0 software. A two-tailed test with statistical significance set at p < 0.05 will be adopted.

ELIGIBILITY:
Inclusion Criteria:

1. The main diagnosis at admission of CHD.
2. Age ≥20 years.
3. Owns an iOS or Android smartphone and can use it.
4. Conscious, clear and can communicate.
5. Agrees to participate in the research after explanation and is willing to use the App.

Exclusion Criteria:

1. Level IV on the New York Heart Association Functional Classification.
2. Left ventricular ejection fraction≦40%.
3. Have a history of severe arrhythmia (e.g., ventricular tachycardia, ventricular fibrillation, complete atrioventricular block).
4. Combined with other serious heart diseases (e.g., congenital heart disease, cardiomyopathy).
5. Mental disorders, end-stage renal disease and other systemic diseases diagnosed by a physician.
6. Severe infection, injury, surgery (e.g., coronary artery bypass graft) or cancer treatment has occurred in the past three months.
7. Physical activities are affected by neurological, respiratory, skeletal, or peripheral vascular diseases.
8. Restricted use of the App due to sensory or cognitive impairment.
9. Already participated in other clinical trials.
10. Planning to receive surgery (e.g., coronary artery bypass graft).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the hospital with a primary diagnosis of CHD will be conducted. We plan to recruit a group of patients to receive the tele-CR program and evaluate the usability of the App perceived by patients at 1 and 3 months after discharge. Therefore, we use the t-test (one sample case) statistical method and set the effect size to a moderate 0.5, power is 0.8, alpha is 0.05 (two-tailed), and the number of samples required after calculation using G*power 3.1 software is 34. Considering the 20% attrition rate, we estimate that we will recruit 45 cases (quantitative). The number of samples for qualitative research is mainly to achieve data saturation, and according to the literature, it is recommended to have at least 12 people.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Level of recruitment rate of tele-CR program | through study completion, an average of 8 months
  The recruitment rate is a percentage calculated by dividing the number of patients who agreed to participate in the study by the number of patients who met the eligibility criteria, which can reflect the interest of CHD patients in participating in the tele-CR program. The recruitment rate is calculated when the number of sample collections of research subjects is completed.
Level of engagement rate of tele-CR program | 1st, 4th, 8th and 12th weeks after discharge
  The degree of actual operation of the App can be used to reflect the degree to engage of the tele-CR program of participants. The researchers collected data on participants' actual use of the App through the App manager's backend, including the number of times knowledge was browsed, the percentage of execution of homework records, and the number of questions asked.
Level of retention rate of tele-CR program | 1st, 4th, 8th and 12th weeks after discharge
  The retention rate refers to the percentage of participants who have not dropped out of the study and can be kept in touch via Line or telephone. It can be used to reflect the extent to which participants remain in the -CR program and help researchers understand the feasibility of future intervention study of the tele-CR program.

SECONDARY OUTCOMES:
Level of acceptance of App and management platform | 4th and 12th weeks after discharge
  The Technology Acceptance Model Scale consists of 11 questions covering three aspects: perceived usefulness, perceived ease of use, and intention to use. Each item is given a score of 1 (strong disagree ) to 7 (strong agree) points respectively. The total score ranges from 11 to 77. The higher the total score of the overall scale, the higher the acceptance of the App.
Level of usability of App and management platform | 4th and 12th weeks after discharge
  The Systems Usability Scale consists of 10 questions, with each question scoring from 1 (strongly disagree) to 5 (strongly agree), including 5 positive questions and 5 negative questions. The total score ranges from 0 to 100 after calculation and conversion. The higher the score, the better the App usability.
Level of satisfaction of App and management platform | 4th and 12th weeks after discharge
  In order to understand the overall satisfaction after using the App, we added a question at the end of the questionnaires: "How do you think your overall satisfaction with using this system is?" The Visual Analogue Scale was used to measure the satisfaction of the user on a 0-10 scale. The higher the score, the higher the overall satisfaction.
Qualitative feedback perception on tele-CR program | 8th weeks after discharge
  The researchers conducted one-on-one semi-structured interviews with participants and evaluated and gained insights into participants' opinions and positive and negative feedback on the App and tele-CR program through thematic content analysis. The interview guidelines are as follows: (1) Please tell us what you think (feel) about participating in this activity over the past three months? (2) Please tell us how you felt when you first started using this App? How do you feel now? (3) What do you think are the conveniences of using this App? What are some of the features you like about it? Why? (4) What inconveniences do you find in using this App? What do you dislike about it? What are the reasons? (5) What suggestions do you have for this App? (6) What suggestions do you have for this entire activity?

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Ching Tsai, Associated Professor, Principal Investigator — Chang Gung University of Science and Technology
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Guishan Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No
The anonymized datasets and study protocols will be available upon reasonable request for academic purposes following the study's conclusion.